CLINICAL TRIAL: NCT01644110
Title: A Phase-Ib/II Study of Ruxolitinib and Pomalidomide Combination Therapy in Patients With Primary and Secondary Myelofibrosis
Brief Title: Ruxolitinib and Pomalidomide Combination Therapy in Patients With Primary and Secondary MF
Acronym: POMINC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Konstanze Doehner, Prof. Dr. Konstanze Doehner, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POMINC(MPNSG02-12); 2012-002431-29 (EudraCT Number)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2023-05

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis; PMF; SMF; Post-PV MF; Post-ET MF
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Intervention Model Description: Cohort 1 (Patient 1 - Patient 41): ruxolitinib treatment will be started at 10 mg twice daily up to 25 mg twice daily, whereas the dose of pomalidomide will be 0.5 mg once daily.
  Cohort 2 (Patient 42 - Patient 90): ruxolitinib treatment will be started at 10 mg twice daily up to 25 mg twice daily, whereas the dose of pomalidomide will be started at 0.5 mg once daily up to 2 mg once daily.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ruxolitinib/pomalidomide (Experimental): Cohort 1 (Patient 1 - Patient 41): ruxolitinib treatment will be started at 10 mg twice daily up to 25 mg twice daily, whereas the dose of pomalidomide will be 0.5 mg once daily.
  Cohort 2 (Patient 42 - Patient 90): ruxolitinib treatment will be started at 10 mg twice daily up to 25 mg twice daily, whereas the dose of pomalidomide will be started at 0.5 mg once daily up to 2 mg once daily.
  Interventions: Drug: INCB018424/CC-4047

INTERVENTIONS:
Drug: INCB018424/CC-4047 — Cohort 1: For patients (1-41) the starting dose of ruxolitinib in this trial is 10 mg twice daily po; pomalidomide will be administered at a permanent dose of 0.5 mg po once daily.
  Cohort 2: For patients (42-90) the starting dose of ruxolitinib in this trial is 10 mg twice daily po; the starting dose of pomalidomide is 0.5 mg po once daily.

SUMMARY:
The proposed study is an open-label, single-arm, Phase-Ib/II trial to assess the efficacy of oral drug combination ruxolitinib and pomalidomide in primary and secondary MF patients.

DETAILED DESCRIPTION:
The proposed study is an open-label, single-arm, Phase-Ib/II trial to assess the efficacy of oral drug combination ruxolitinib and pomalidomide in primary and secondary MF patients. Dosages of the drugs are derived from previous Phase-I/II studies; ruxolitinib treatment will be started at 10 mg twice daily, whereas the dose of pomalidomide will be 0.5 mg once daily.

Dose reductions and discontinuations will be allowed in case of myelosuppressive effects.

Intra-patient dose escalation will be permitted for ruxolitinib to optimize efficacy of the therapeutic regimen; pomalidomide will be given in a permanent dosage of 0.5mg per day.

Treatment response will be evaluated continuously after each treatment cycle (1 cycle = 28 days) according to the IWG-MRT criteria expanded by the response criterion RCT-independency.

In case of progressive disease study therapy will be stopped; In patients showing response or stable disease, continuous therapy within the study is intended for a maximum of 12 treatment cycles; After completion of 12 treatment cycles, therapy can be continued if a measurable benefit of treatment is evident. This extension has to be discussed between the local and the principle investigator. Conditions leading to patient withdrawal from the study are detailed in the protocol "PATIENT WITHDRAWAL FROM STUDY PARTICIPATION".

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of voluntarily signing an IRB/IEC-approved informed consent
2. Diagnosis of Myeloproliferative Neoplasms (MPN) either de novo myelofibrosis according to current WHO criteria (PMF), secondary myelofibrosis (post-PV MF and post-ET MF) according to the IWG-MRT consensus terminology) (Appendix I)
3. Anemia with hemoglobin level of <10 g/dl or transfusion-dependent anemia*
4. Splenomegaly (>11 cm total diameter) and/or leukoerythroblastosis
5. Adequate organ function, i.e. ALT and/or AST <3 x upper limit of normal (ULN), total bilirubin <3 x ULN, and serum creatinine <2 mg/dl
6. Subject must be willing to receive transfusion of blood products
7. ECOG performance status <3
8. Females of childbearing potential (FCBP) must undergo repetitive pregnancy testing (serum or urine) and pregnancy results must be negative.**
9. Reliable contraception should be maintained throughout the study and for 28 days after study treatment discontinuation*
10. Unless practicing complete abstinence from heterosexual intercourse, sexually active FCBP must agree to use adequate contraceptive methods*
11. Males (including those who have had a vasectomy) must use barrier contraception (condoms) when engaging in sexual activity with FCBP. Males must agree not to donate semen or sperm*
12. All subjects must:

    * understand that the investigational product could have a potential teratogenic risk.
    * be counseled about pregnancy precautions and risks of fetal exposure.
    * agree to abstain from donating blood while taking investigational product.
    * agree not to share study medication with another person and to return all unused study drug to the investigator.

Exclusion Criteria:

1. Patients eligible for hematopoietic stem cell transplantation (suitable candidate and suitable donor is available)
2. Patients with response to standard therapy as recommended by the Deutsche Gesellschaft für Hämatologie und Medizinische Onkologie (DGHO/Onkopedia)
3. Pregnant or breast feeding females
4. BCR/ABL-positivity
5. Diagnosis of ET (according to WHO 2016 criteria)
6. Diagnosis of PV (according to WHO 2016 criteria)
7. >20% blasts in peripheral blood or bone marrow
8. thrombocytopenia <100 /nl or transfusion-dependent thrombocytopenia
9. neutropenia <0.5 /nl
10. Known positive status for HIV, HBV or HCV
11. Prior treatment with IMiDs (thalidomide, lenalidomide, pomalidomide) or with Interferon-alpha within a 3 month time period before Screening-phase
12. Patient treatment with Ruxolitinib within a 14 days time period before Screening-phase
13. History of thrombosis or pulmonary embolism within 6 months prior to study entry
14. Peripheral neuropathy >grade 1 CTC
15. No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician about study participation.
16. Presence of any medical/psychiatric condition or laboratory abnormalities which may limit full compliance with the study, increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study
17. Drug or alcohol abuse within the last 6 months
18. History of malignancy except for i) adequately treated local basal cell or squamous cell carcinoma of the skin, ii) asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to randomization, or iii) any other cancer that has been in complete remission for ≥ 5 years
19. Patients undergoing treatment with hematopoietic growth factor receptor agonists (i.e., erythropoietin [Epo], granulocyte colony stimulating factor (GCSF [Neupogen; Neulasta], romiplostim, eltrombopag) within a 4 weeks period prior to screening-phase.
20. Patients receiving any medication listed in the Appendix V "Prohibited Medications" (within 7 days prior to the first dose of study drug).
21. Patients with clinically significant bacterial, fungal, parasitic or viral infection which require therapy. Patients with acute bacterial infections requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed.
22. Patients under ongoing treatment with another investigational medication or having been treated with an investigational medication within 28 days of screening.
23. No consent for biobanking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-08; Primary Completion 2024-04 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Best response rate within 12 treatment cycles according to the IWG-MRT criteria (including CR, PR, CI) and red cell transfusion (RCT) independency according to Gale et al 2010 and 2011). | one year
  Best response rate within 12 treatment cycles according to the IWG-MRT

SECONDARY OUTCOMES:
Overall safety profile of ruxolitinib and pomalidomide combination observed during treatment, as well as cumulative incidence of leukemic transformation | one year
  Overall safety profile of ruxolitinib and pomalidomide combination characterized by type, frequency, severity (graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 3.0), timing and relatedness of adverse events (AEs) and laboratory abnormalities observed during treatment, as well as cumulative incidence of leukemic transformation
Progression-free survival | three years
  Progression-free survival
duration of response | three years
  duration of response
overall survival | three years
  overall survival
Quality of life assessed by the Myeloproliferative Neoplasm Symptom | three years
  Quality of life assessed by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF Protocol 5/25/11), change in ECOG performance status from study entry to each visit where the variable is measured.
Clinical Benefit - Assessment of each patient | three years
  Clinical Benefit:
  * Lab / Clinical data: Stable disease (SD) plus hematologic improvement: prolongation of RBC transfusion intervals by ≥50% compared to baseline in transfusion dependent patients or ≥1 g/dL Hb increase in the absence of RBC transfusion dependency and/or
  * Questionaire: Stable disease (SD) plus improvement of MF-associated symptoms: SD plus improvement of at least one MF-associated symptom according to the MPN-SAF / EORTC QLQ-C30 or FACT-Lym by a minimum of 50% and/or SD plus improvement of ≥ two MF-associated symptoms according the MPN-SAF / EORTC QLQ-C30 or FACT-Lym by a minimum of 25% each.
Monthly Response assessment | three years
  Response criteria:
  Assessment according to the IWG-MRT (based on lab, clinical data): CR / PR / CI / PD / SD / RD/ RBC-TD / RBC-TI

CONTACTS AND LOCATIONS:
Overall Officials: Konstanz Doehner, MD, Principal Investigator — University of Ulm
Locations (17):
- Germany (17):
  - Universitätsklinikum Aachen - Med. Klinik IV, Aachen
  - Hämatologisch onkologische Praxis, Augsburg
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Klinik für Innere Medizin Uniklinik Köln, Cologne
  - BAG Freiberg-Richter, Jacobasch, Wolf, Illmer, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Uniklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Universitätsklinikum Tübingen, Tübingen
  - University of Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No